CLINICAL TRIAL: NCT04068558
Title: Synchronized Nasal Intermittent Positive Pressure Ventilation Versus Noninvasive Neurally Adjusted Ventilatory Assist Ventilation in Extremely Premature Infants: a Randomized Crossover Trial
Brief Title: sNIPPV Versus NIV-NAVA in Extremely Premature Infants
Acronym: EASYNNEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EASYNNEO; 2019-A00420-57 (Other: ID-RCB)
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Premature Birth; Ventilator Lung; Newborn
Keywords: neurally adjusted ventilatory assist; synchronized nasal intermittent positive pressure ventilation
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: Randomized crossover trial in the Neonatal Intensive Care Unit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VNI-NAVA/sNIPPV (Experimental): Ventilation of the child non-invasive ventilation (VNI) NAVA then sNIPPV
  Interventions: Device: VNI-NAVA/sNIPPV
- sNIPPV/VNI-NAVA (Experimental): Ventilation of the child sNIPPV then non-invasive ventilation (VNI) NAVA
  Interventions: Device: sNIPPV/VNI-NAVA

INTERVENTIONS:
Device: VNI-NAVA/sNIPPV — Ventilation of the child in NIV-NAVA for 2 hours then ventilation of the child in sNIPPV for two hours. The ventilation periods consist of one hour of wash-out and one hour of data collection
  Arms: VNI-NAVA/sNIPPV
Device: sNIPPV/VNI-NAVA — Ventilation of the child in sNIPPV for 2 hours then ventilation of the child in NIV-NAVA for two hours. The ventilation periods consist of one hour of wash-out and one hour of data collection
  Arms: sNIPPV/VNI-NAVA

SUMMARY:
The aim of this study is to demonstrate a significant decrease in asynchrony with NIV-NAVA using the Servo n ventilator (Getinge, Sweden), as compared to abdominal triggered (Graseby capsule) synchronized nasal intermittent positive pressure ventilation (sNIPPV) using the Infant Flow CPAP device (Care Fusion, USA).

All of the data obtained can be used to develop a large-scale study aimed at reducing the rate of re-intubation in the study population (pilot study). In fact, the re-intubation criteria for extremely premature children are based on clinical criteria (desaturations, apnea, signs of respiratory control) and paraclinical criteria (FiO2, Potential hydrogen (pH), PCO2).

The results of this pilot study will help to develop an adapted methodology and to calculate a sample size to compare the 2 modes of NIV to the test on a clinical criterion: the rate of re-intubation after extubation, which is classically high in these patients.

DETAILED DESCRIPTION:
The use of non-invasive ventilation has significantly reduced morbidity and mortality in premature newborns by reducing the pulmonary lesions caused by invasive ventilation. Currently, variable flow continuous positive airway pressure (CPAP) devices, such as the infant flow® driver, are considered more efficient than constant flow pressure sources. Nasal intermittent positive pressure ventilation, as compared to CPAP, might reduce the extubation failure rate, but has no impact on mortality or bronchopulmonary dysplasia. However, data is lacking on the interest of synchronization and on the effect of the different available interfaces (prongs, masks, cannulas). In addition, the ventilatory characteristics (high respiratory rate and low inspiratory effort) of the premature infant increase the risk of asynchrony between the patient and the ventilator, which is a major cause of poor tolerance for this type of ventilation.

NAVA (neurally adjusted ventilatory assist) is a recent ventilatory mode that offers proportional assistance to respiratory work based on the measured electrical activity of the diaphragm via oesophageal electrodes. It thus allows a regulation of inspiratory pressures and time by the patient him/herself. The physiological effects of NAVA have been primarily described in intubated neonates and studies have shown a significantly improved synchronization and significantly decreased inspiratory pressures in patients ventilated with NAVA compared to intermittent controlled ventilatory support. However, the currently available evidence is limited and no beneficial effect on morbidity or mortality has been identified so far .

There are few studies on noninvasive NAVA (NIV-NAVA) conducted exclusively in neonates, most of which included a limited number of patients. Only one study to date compared NIV-NAVA to another synchronized NIV mode (NIV pressure support) using the Servo-i ventilator. This prospective crossover study found a significant decrease in peak inspiratory pressure (PIP), FiO2, frequency and length of desaturations in the NIV-NAVA group.

Decreased asynchrony has been observed during NIV-NAVA as compared to pressure-support NIV In adult patients and in 6 children hospitalized in the Pediatric ICU (median age 18 months).

In premature neonates, variable flow CPAP is preferentially used. Synchronized intermittent positive pressure can be delivered using a variable flow device and a Graseby abdominal capsule. Since variable flow CPAP is considered the most efficient pressure generator, it is legitimate to compare synchronization performance of the variable flow synchronized nasal intermittent positive pressure ventilation (sNIPPV) to NIV-NAVA. This comparison has never been performed so far, to our knowledge.

We hypothesize that synchronization will be markedly improved with NIV-NAVA as compared to sNIPPV.

ELIGIBILITY:
Inclusion criteria:

* Premature infants born before 28 weeks of gestation
* Corrected age below 32 weeks of gestation
* Postnatal age > or = 3 days
* Receiving NIPPV (any mode)
* Equipped with an Edi catheter
* Receiving caffein treatment
* Parental consent
* Recipient of French social security coverage

Non-inclusion criteria:

* More than 1 apnea/hour requiring bag-mask ventilation, or pH<7.2 and/or TcPCO2>70, or FiO2>0.6 in the previous 6 hours.
* Nasal trauma precluding the use of non-invasive ventilation
* Major congenital anomalies
* Grade III or higher intraventricular hemorrhage
* Use of anesthetics or sedative within the past 24 hours, except opioids for iatrogenic withdrawal treatment
* Hemodynamic compromise defined as a mean blood pressure less than gestational age (in mmHg) or a capillary refill time more than 3 seconds
* Neuro-muscular disorders

Min Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Asynchrony index | 4 hours
  Asynchrony index as previously defined in the literature using the following parameters: Ineffective effort (IE): presence of an inspiratory electromyographic signal not followed by pressurization; Late cycling (LC): a cycle with an inspiratory time greater than twice the patient's neural inspiratory time; Premature cycling (PC): a cycle with an inspiratory time shorter than the the neural inspiratory time; Double triggering (DT): two ventilator-delivered cycles triggered by one neural inspiration; Auto triggering (AT): a cycle delivered by the ventilator in the absence of EAdi signal.

SECONDARY OUTCOMES:
Components of the Asynchrony index | 4 hours
  Each component of the Asynchrony index will be compared between the 2 ventilatory modes.
Mean change in electric activity of the diaphragm (Edi) | 4 hours
  Analyze as exploratory data of Mean delta Edi (max-min value) in NIV NAVA vs sNIPPV
Apnoea | 4 hours
  Analyze as exploratory data of Frequency of apnoea
Desaturations | 4 hours
  Analyze as exploratory data of Frequency of desaturations below 80%
Bradycardia | 4 hours
  Analyze as exploratory data of Frequency of bradycardia < 100 bpm
ComfortNeo score | 4 hours
  Analyze as exploratory data of Comfort Neo score assessed by the nurse before and after each ventilation period
transcutaneous PCO2 | 4 hours
  TcPCO2 modeling over time and comparison between NIV Nava and sNIPPV
Nava level | 1 hour
  Description of Nava levels used during NIV Nava
Inspiratory pressure during sNIPPV | 1 hour
  Description of inspiratory pressures used during sNIPPV
Bag-mask ventilation or re-intubation | 4 hours
  Frequency of bag-mask ventilation or re-intubation
Re-intubation within 7 days | 7 days
  Frequency of re-intubation within 7 days of randomization
Fi02 | 4 hours
  FiO2 changes over time during NIV NAVA and sNIPPV

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No